CLINICAL TRIAL: NCT06155357
Title: Pre-habilitation Multicomponent Lifestyle Program for Patients Undergoing Ablation for Atrial Fibrillation
Brief Title: A Study of a Lifestyle Program on Recurrent Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda R. Bonikowske, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-003042
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Interventions Pre-Procedure (Experimental): Subjects with paroxysmal or persistent atrial fibrillation (AF) who are scheduled to undergo elective catheter ablation of AF will participate in a 12-week multicomponent lifestyle intervention program.
  Interventions: Behavioral: Multicomponent lifestyle intervention program
- Standard of Care (No Intervention): Subjects who have previously undergone catheter ablation of atrial fibrillation (AF) as part of their standard of care will have medical chart review completed to gather information.

INTERVENTIONS:
Behavioral: Multicomponent lifestyle intervention program — The multicomponent lifestyle intervention program is targeted at risk factor management, increased exercise capacity, and weight loss. The program will commence upon order/referral for ablation. Ablation would occur during the lifestyle program and the program will be continued after the ablation to complete 12 weeks or up to 36 exercise sessions.
  Arms: Lifestyle Interventions Pre-Procedure

SUMMARY:
The purpose of this study is to examine the impact of a comprehensive lifestyle intervention, including cardiac rehabilitation, prior to catheter ablation (a procedure to stop abnormal electrical signals in the heart), on Atrial Fibrillation (AF)-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation.
* Planned elective catheter ablation of AF.

Exclusion Criteria:

* Prior catheter ablation.
* Presence of pacemaker/ICD.
* Longstanding persistent AF.
* Uncontrolled AF (including poor rate control or tachycardia-mediated cardiomyopathy requiring urgent cardioversion/ablation at the clinician's assessment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Cardiac Rehab Sessions Attended | 12 weeks
  Number of cardiac rehab sessions attended during the 12-week multicomponent lifestyle intervention program.

SECONDARY OUTCOMES:
Number of subjects with Atrial Fibrillation (AF) recurrence | 1 year
  Number of subjects with AF recurrence will be assessed by chart review and clinically indicated holter monitor.
Change in weight loss | Baseline, 12 weeks
  Change in weight loss pre & post multicomponent lifestyle intervention program reported in kilograms (kg)
Change in exercise capacity | Baseline, 12 weeks
  Change in exercise capacity will be assessed by 6-minute walk test pre & post multicomponent lifestyle intervention program. Measurement (meters) of distance a person can walk on flat ground in 6 minutes.
Change in Atrial Fibrillation (AF) Symptom severity | Baseline, 12 weeks, 6 months, 1 year
  Change in AF Symptom Severity will be assessed by the Atrial Fibrillation Severity Scale (AFSS) questionnaire. The AFSS questionnaire is a 19-item self-administered questionnaire developed to capture subjective and objective ratings of AF related symptoms, health care utilization, and AF disease burden, including frequency, duration, and severity of episodes. Higher scores indicate higher symptom severity (range of 0-35).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bonikowske, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials